CLINICAL TRIAL: NCT07296770
Title: An Artificial Intelligence Driven Approach to Optimize Patient Selection for a Transitional Pain Service
Acronym: TPS-Select
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-42631
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Postsurgical Pain Management; Postsurgical Pain, Chronic; Opioid Use After Surgery
Keywords: Pain; Transitional Pain Service; Postsurgical Pain; Postoperative Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Oxycodone; Hydrocodone; Acetaminophen; Morphine; Methadone; Buprenorphine; Gabapentin; Duloxetine Hydrochloride; Pregabalin; Amitriptyline; Nortriptyline; Acupuncture Therapy; Injections, Intra-Articular; Radiofrequency Ablation; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: After a patient joins the study, they will be randomly assigned to either the standard care group or the Transitional Pain Service (TPS) group. The assignment will be done by the study coordinator using a process that makes sure patients are evenly matched based on their level of risk. All patients in the study are considered high-risk, but the investigators will sort them into three groups-mildly severe, moderately severe, and extremely severe-to help ensure that similar patients are compared fairly across both study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Transitional Pain Service (Experimental): Patients assigned to the Transitional Pain Service group will receive extra support before and after surgery to help with pain and recovery. This may include educational videos, meetings with a pain pharmacist for safe medication use and tapering, mental health screening with referrals to supportive resources, and physical therapy. Patients may also be offered pain-relief procedures or treatments such as nerve blocks, injections, imaging, or other outpatient therapies provided by pain specialists. These services are meant to support recovery, and patients may choose how much to participate while remaining in the study even if all activities are not completed.
  Interventions: Device: TPS-Select; Drug: Pharmacologic Pain Management; Procedure: Interventional Pain Procedures; Behavioral: Psychological Management and Pain Education; Behavioral: Physical Therapy
- Usual Care (No Intervention): In this arm, patients will receive usual surgical care. However, patients will still complete the questionnaires and will also have the option of a pharmacist wellness check-in at 60 days after surgery.

INTERVENTIONS:
Device: TPS-Select — TPS-Select is a computer-based tool that helps the research team identify patients who may be eligible for this study. It uses information that already exists in the medical record at the time a surgery is scheduled to estimate the chance of developing ongoing pain after surgery. This information can include details about the planned surgery, prior medical conditions, past surgeries, and previous use of pain medications.
  The tool runs automatically and is used only to help the research team decide whom to contact about possible participation in the study. The risk estimate created by this tool is not added to the medical record and is not seen by the patient's care team. Only approved members of the research team can see this information through a secure research system.
  Arms: Transitional Pain Service
Drug: Pharmacologic Pain Management — A pharmacist will meet with patients as part of the Transitional Pain Service before and after surgery. During this visit, the pharmacist will work with patients to create a personalized pain management plan, using the medications stated in this intervention to help safely and effectively control pain. This will guide patients on the proper use of opioid analgesics and non-opioid analgesics, including acetaminophen, non-steroid anti-inflammatory drugs, gabapentinoids, and topical medications to manage surgical pain.
  Other Names: Oxycodone Hydrochloride; Hydrocodone Bitartrate and Acetaminophen; Morphine Sulfate; Methadone Hydrochloride; Buprenorphine; Gabapentin; Duloxetine Hydrochloride; Pregabalin; Amitriptyline Hydrochloride; Nortriptyline Hydrochloride
  Arms: Transitional Pain Service
Procedure: Interventional Pain Procedures — If a patient has significant pain after their surgery, the care team may evaluate the patient for additional pain-relief options, such as the interventional pain procedures listed above. Local numbing medication or imaging studies may also be used to ensure the treatment is safe and appropriate. All anesthesiologists on the pain service are specially trained to perform these procedures. Only approved procedures will be offered, along with any imaging needed for evaluation.
  Other Names: Epidural Steroid Injection; Acupuncture; Trigger Point Injection; Peripheral Nerve Block; Joint Injection; Radiofrequency Ablation
  Arms: Transitional Pain Service
Behavioral: Psychological Management and Pain Education — Patients will be asked to complete short online pain education modules to help set expectations and prepare for pain after surgery. These materials are available at https://www.transitionalpainservice.ca/learn. Each patient will also be screened for mood-related concerns, including symptoms of depression, using a brief questionnaire. If a patient has significant symptoms of depression, they may be referred to a pain psychologist and, if needed, a UCSF psychiatrist for additional support. These visits may include proven approaches such as cognitive behavioral therapy, acceptance and commitment therapy, and mindfulness-based strategies to help patients manage pain, cope with stress, and improve daily functioning. Patients with milder symptoms may be referred to group-based pain psychology sessions led by a pain psychologist.
  Arms: Transitional Pain Service
Behavioral: Physical Therapy — Patients will be assessed for their physical function and ability to carry out daily activities. If a patient has difficulty with mobility, strength, or endurance, they may be referred to physical or occupational therapy before surgery to help improve overall conditioning. Pre-surgery therapy may include exercises to strengthen the core, arms, and legs, improve balance, and build stamina, as well as an overall fitness assessment. Referrals will only be made if it is safe for the patient to participate, and standard safety checks-such as heart health and fall risk-will be completed beforehand. All therapy will be provided by a licensed physical therapist using established, evidence-based treatment plans.
  Arms: Transitional Pain Service

SUMMARY:
The goal of this clinical trial is to learn whether a pain-management program called a Transitional Pain Service can help prevent long-term pain and reduce opioid needs after surgery in adult surgical patients who may be at higher risk for developing persistent pain. The main questions this trial aims to answer are: 1) Does the Transitional Pain Service help high-risk surgical patients manage pain better after surgery? 2) Can a computer tool (an algorithm) improve screening of patients for long-lasting pain after surgery? The investigators will compare patients who continue with their usual care to patients who receive support from the Transitional Pain Service to see if the program leads to better pain control and lower opioid use. Participants will share information about their pain levels and the pain-relief treatments they are using before and after surgery so researchers can better understand how the program affects recovery. Patients assigned to the Transitional Pain Service will also be offered additional coordinated support before and after their surgery to help optimize their pain control and overall recovery.

ELIGIBILITY:
Patients may take part in this study if they:

* Are 18 years or older
* Are having a planned (elective) surgery at UCSF
* Are identified as higher risk for chronic pain after surgery by a computer model
* Agree to join the study and sign consent

Patients cannot take part if they:

* Have too much missing information in their medical record (more than 75%)
* Have a surgery scheduled less than 1 month away
* Have serious memory or thinking problems that make participation difficult
* Are in another clinical study that would interfere with this one
* Do not live in California
* Choose not to participate or sign consent
* Have severe depression with suicidal thoughts that requires urgent care
* Are pregnant or breastfeeding

A patient who has already joined may be removed from the study if they:

* Cannot complete most of the scheduled follow-up phone calls or pre-surgery recommendations (up to 6 months after discharge)
* Pass away between the surgery booking date and 6 months after leaving the hospital
* Become pregnant in the 6 months after discharge

Patients may remain enrolled but their data may not be used in the main study results if they experience:

* A long-lasting infection after surgery
* Hardware problems related to their surgery (for example, issues with implanted devices)
* A major injury or life event that affects their pain levels, such as a significant fall or an emergency surgery
* Difficulty completing the planned follow-up phone calls up to 6 months after discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients With Chronic Post-Surgical Pain | 90 days after date of surgery
  This outcome measures how many patients in each group (Standard of Care vs. Transitional Pain Service) have chronic post-surgical pain 90 days after date of surgery. Chronic post-surgical pain refers to pain that starts after surgery and lasts longer than 3 months, gets worse after 3 months, or spreads to nearby nerves or areas connected to the surgical site. To make this diagnosis, other causes-such as infection, cancer, or pain conditions from before surgery-must be ruled out.

SECONDARY OUTCOMES:
Opioid Use After Surgery | 30, 60, and 90 days after discharge from hospital
  This measures the amount of opioid medication patients are using after surgery, recorded as morphine milligram equivalents (MMEs). Average MMEs will be compared between groups to see whether the program helps reduce opioid needs.
Pain Levels After Surgery | 30, 60, and 90 days after discharge from the hospital
  This outcome looks at patients' reported pain scores over time. The study will compare average pain levels between the two groups to understand how the program affects recovery.
Healthcare Costs | 30, 60, and 90 days after discharge from the hospital
  This measures costs to the hospital related to pain care and recovery after surgery. Average costs will be compared between groups to evaluate whether the Transitional Pain Service may reduce overall costs.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bishara, MD, Principal Investigator — UCSF Department of Anesthesia
Locations (1):
- UCSF Hospitals, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with outside researchers because the information collected in this study includes sensitive health details that could pose privacy risks if shared. Although all data are protected and stored securely, sharing IPD outside the study team may increase the chance of re-identification. To protect patient privacy, only summarized results that do not identify any individual will be shared publicly.